CLINICAL TRIAL: NCT00930696
Title: Extensive Abdominal Lavage Following Laparoscopic Full Thickness Resection of Deep Endometriosis Involving the Bowel, Effects on Post-Operative Inflammation: a Randomised Controlled Trial
Brief Title: Effects of Extensive Abdominal Lavage on Postoperative Inflammation Following Full Thickness Excision of Deep Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Koninckx Philippe, UZ Gasthuisberg, Catholic University Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: trial_lavage_01/endometriosis
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Endometriosis
Keywords: endometriosis; abdominal lavage; bowel perforation; discoid resection; laparoscopy
MeSH Terms: conditions — Endometriosis; Intestinal Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extensive Abdominal Lavage (Experimental): women with full thickness excision of deep endometriosis involving the bowel
  Interventions: Procedure: Extensive abdominal lavage
- Standard Rinsing (Active Comparator): women with full thickness excision of deep endometriosis involving the bowel
  Interventions: Procedure: Rinsing of the abdomen

INTERVENTIONS:
Procedure: Extensive abdominal lavage — Extensive lavage of the abdomen with 8 liters of saline at the end of the surgical procedure
  Arms: Extensive Abdominal Lavage
Procedure: Rinsing of the abdomen — Standard rinsing of the abdomen with some 0,5 liters of saline at the end of the surgical procedure
  Arms: Standard Rinsing

SUMMARY:
Surgical treatment of deep endometriosis with bowel involvement is widely accepted to require complete excision of all endometriosis also when invading the bowel. In case of opening of the bowel a subsequent inflammatory reaction follows the surgery, as demonstrated by the increase in blood levels of C-reactive protein during the first post-operative week. Furthermore it increases the risk of post-operative bowel complications. In case of peritonitis the general surgeons use extensive lavage in order to decreases mortality, morbidity and post-operative adhesions formation, as demonstrated in animal models and clinically in patients with peritonitis. Considering the efficacy of extensive lavage for peritonitis and the inflammatory reaction as judged by the increased C-reactive protein (CRP) following full thickness deep endometriosis resection from the bowel, the study aims to evaluate, in women undergoing this procedure, the effect of extensive abdominal lavage on abdominal inflammation and post-operative bowel complications.

DETAILED DESCRIPTION:
In a consecutive series 20 women with full thickness resection for deep endometriosis received randomly, at the end of the procedure, a standard abdominal rinsing (n=10) or extensive abdominal lavage with 8 Liters of saline (n=10). C-reactive protein and white blood cell count values were collected daily for 7 days. Women were observed for complications during the first post-operative week and during the follow up at 1 and 6 months.

The primary end point was to evaluate the effects of extensive abdominal lavage on post-operative inflammation. Secondary end-point was to explore the potential protective rule against post-operative bowel complications.

ELIGIBILITY:
Inclusion Criteria:

* The patients (aged 18-50 years) were all recruited from a single, tertiary referral hospital at Leuven University, Belgium, specializing in the surgical treatment of severe endometriosis.
* All the women were scheduled for a surgical excision of a rectovaginal nodule.
* Women with a full thickness involvement of the bowel requiring discoid resection were included.

Exclusion Criteria:

* evidence on chest x-ray in the previous 3 months of old or currently active TB, even if adequately treated;
* evidence of serious infections (such as pneumonia or pyelonephritis) in the previous 3 months
* evidence of a documented HIV infection, active hepatitis-B or C, or an opportunistic infection (e.g. herpes zoster, cytomegalovirus, pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) in the previous 6 months
* Previous transplant surgery, a lymphoproliferative disorder or other malignancy
* Positive cervical cytology in the previous 6 months
* Any haematological or biochemical abnormalities on routine screening.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Post-operative C-reactive protein blood values | Daily for 1 week

SECONDARY OUTCOMES:
Bowel complications rate | By the clinicians during the first post-operative week and at 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe R Koninckx, MD, PhD, Principal Investigator — Catholic University Leuven
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Adam U, Ledwon D, Hopt UT. [Programmed lavage as a basic principle in therapy of diffuse peritonitis]. Langenbecks Arch Chir. 1997;382(4 Suppl 1):S18-21. doi: 10.1007/pl00014638. German. PMID 9333702
- [Background] Arnesjo B, Breland U, Petersson BG. The effect of peritoneal lavage on the postoperative course after colonic anastomosis and perforation in the rat. Acta Chir Scand. 1975;141(5):433-6. PMID 1181805
- [Background] Koninckx PR, Timmermans B, Meuleman C, Penninckx F. Complications of CO2-laser endoscopic excision of deep endometriosis. Hum Reprod. 1996 Oct;11(10):2263-8. doi: 10.1093/oxfordjournals.humrep.a019087. PMID 8943540
- [Background] Polubinska A, Winckiewicz M, Staniszewski R, Breborowicz A, Oreopoulos DG. Time to reconsider saline as the ideal rinsing solution during abdominal surgery. Am J Surg. 2006 Sep;192(3):281-5. doi: 10.1016/j.amjsurg.2005.05.047. PMID 16920418
- [Background] Ret Davalos ML, De Cicco C, D'Hoore A, De Decker B, Koninckx PR. Outcome after rectum or sigmoid resection: a review for gynecologists. J Minim Invasive Gynecol. 2007 Jan-Feb;14(1):33-8. doi: 10.1016/j.jmig.2006.07.015. PMID 17218226
- [Background] Sortini D, Feo CV, Maravegias K, Carcoforo P, Pozza E, Liboni A, Sortini A. Role of peritoneal lavage in adhesion formation and survival rate in rats: an experimental study. J Invest Surg. 2006 Sep-Oct;19(5):291-7. doi: 10.1080/08941930600889409. PMID 16966207